CLINICAL TRIAL: NCT06410196
Title: Modulating Explore-exploit Biases by Improving Mood in Adults With Methamphetamine Use Disorder
Brief Title: Mood and Decision-making in Methamphetamine Use Disorder
Acronym: MDM-MUD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Laureate Institute for Brain Research, Inc. (Other)
Collaborators: National Institute of General Medical Sciences (NIGMS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 2024-002; P20GM121312 (NIH)
Record Dates: First submitted 2024-05-03; First posted 2024-05-13 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-09

CONDITIONS: Methamphetamine Abuse

STUDY DESIGN:
Intervention Model Description: 80 participants to be enrolled in the study, with 40 in each arm (randomized arm allocation)
Who Masked: Participant, Investigator
Masking Description: At the beginning of the study, the participants and experimenter are blind to the arm allocation. The experimenter's blindness is lifted upon administering the intervention while the participant's blindness is maintained until the end of their participation in the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Positive mood modulation (Active Comparator): Use of happy/positive autobiographical memories which are vivid, emotionally pleasurable and not drug-related, as assessed by individual interview and ratings
  Interventions: Behavioral: Mood modulation
- Neutral mood modulation (Sham Comparator): Use of neutral/procedural autobiographical memories which are vivid, emotionally neutral and not drug-related, as assessed by individual interview and ratings
  Interventions: Behavioral: Mood modulation

INTERVENTIONS:
Behavioral: Mood modulation — Autobiographical memory recall designed to modulate mood and affective state by reminiscing about personal life events
  Other Names: Autobiographical memory recall

SUMMARY:
In this project, the investigators examine behavior and associated brain activity during explore-exploit decision-making tasks performed pre- and post-modulation of affective state using autobiographical memory recall. The investigators hypothesize that a positive memory recall will reduce negative affective state, reduce explore-exploit biases and normalize the associated brain activity. The investigators propose a randomized double-blind, sham-controlled trial of positive autobiographical memory recall with 80 adults (n=40 per arm) with methamphetamine use disorder (MUD) currently involved in abstinence only treatment centers.

DETAILED DESCRIPTION:
The growing epidemic of methamphetamine use disorder (MUD) is a significant burden on public health with surging overdose deaths, high likelihood of relapse, and current lack of approved medication to treat the disorder. When it comes to decision-making, individuals with MUD often prioritize drug over non-drug rewards despite negative life consequences; in addition, they may not sufficiently "explore" all available choices to "exploit" the best one (in other words, make the optimal choice leading to positive consequences). Therefore, the "explore-exploit" trade-off is often dysfunctional in MUD. Decision-making imbalances in the explore-exploit trade-off may extend well into abstinence, a period marked by a negative affective state (low mood, high depression and anxiety, withdrawal), which in turn triggers heightened craving and subsequent drug use urges. The insula, anterior cingulate cortex and striatum are crucial brain regions involved in explore-exploit behaviors and affective state signaling that have also been linked to drug reward processing in MUD. We propose that reducing negative affective state (improving mood) could help normalize explore-exploit behaviors and the response of these brain areas in individuals currently abstinent from methamphetamine and other drugs. This project will use a non-drug-related autobiographical memory recall to improve the mood of individuals with MUD and measure whether it normalizes non-drug decision-making, using a functional magnetic resonance imaging-based 3-arm bandit task and a behavioral contextual reinforcement learning task. A mixed experimental design in n=80 (72 completers, assuming 10% attrition) allows the identification of a between-subjects effect of positive (n=40, 36 completers) vs. neutral (n=40, 36 completers) mood modulation and assess the within-subject impact on explore-exploit behaviors pre- versus post-mood modulation. Mood groups will be compared on positive and negative affect, and behavioral/brain responses to reward valuation, outcomes and learning rates.

The overarching goal is to establish that improving mood in individuals with MUD can reduce their negative affective state, normalize outcome sensitivity in key brain regions and associated learning, and reduce the influence of drug rewards on the valuation of non-drug rewards. This approach of this proposal embodies the goals of the NIH RDoC Initiative and the NeuroMAP Center by identifying an actionable disease-modifying target (mood) and studying its effect on the cognitive and neural dysfunction underlying a specific cognitive process (explore-exploit behaviors) relevant to MUD, and possibly other related neuropsychiatric disorders. By targeting the intertwined mechanisms between negative affect and explore-exploit biases, innovative, effective intervention strategies for MUD may be unveiled, addressing a critical public health challenge.

ELIGIBILITY:
Inclusion Criteria:

* Adults 18-65 years old
* English proficiency as evaluated by language ability during screening
* Past-year diagnosis of DSM-5 methamphetamine use disorder (MUD) confirmed by the MINI
* Actively enrolled in treatment for substance use disorder.

Exclusion Criteria:

* Severe traumatic brain injury (as indicated by a score ≥3 on the Tulsa Head Injury Screen
* Any medical condition interfering with the participation in the study as determined by medical screening
* DSM-5 diagnosis of psychotic disorders, bipolar I disorder, or major depressive disorder with psychosis
* fMRI contraindications as listed on the MR environment screening form
* Positive breathalyzer for alcohol
* Positive urine drug screening, except for cannabis or prescribed benzodiazepines, as indicated in the medical screening
* Evidence of inability to comply with study procedures based on judgement of the experimenter.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-07-26 (Actual); Primary Completion 2027-07-01 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
Current affective state | Change from pre-intervention (baseline) to post-intervention (90min later) on study day 1
  Use of PANAS-PA and PANAS-NA questionnaires to measure positive and negative affect respectively (scale range: 0=low; 60=high; low mood is defined as low positive and/or high negative affect)
Learning rates | Change from pre-intervention (baseline) to post-intervention (30min later) on study day 1
  Computational modeling is used to compute how fast (learning rate) participants update their choice strategy following appetitive and aversive outcomes during 3-arm bandit task
Response to punishment in insular cortex | Change from pre-intervention (baseline) to post-intervention (30min later) on study day 1
  BOLD signal is used to measure the activity in the insula as a predefined region of interest (ROI), using Brainnetome atlas, following the delivery of aversive outcomes during 3-arm bandit task
Correct choice rate of mid-value option in contexts 1 (M1) and 2 (M2) during the testing phase | Change from pre-intervention (baseline) to post-intervention (60min later) on study day 1
  Proportion of trials for which the mid-value option is correctly chosen when paired against a high- or low-value option during contextual RL task
∆BIC for absolute vs. relative value coding | Change from pre-intervention (baseline) to post-intervention (60min later) on study day 1
  Difference in model-fitting between the absolute and intrinsically enhanced or range adaptive (relative) models as measured by Bayesian Information Criterion (∆BIC) during contextual RL task

SECONDARY OUTCOMES:
Response to punishment in anterior cingulate cortex (ACC) | Change from pre-intervention (baseline) to post-intervention (30min later) on study day 1
  BOLD signal is used to measure the activity in the ACC as a predefined ROI, using Brainnetome atlas, following the delivery of aversive outcomes during 3-arm bandit task
Response to punishment in striatum | Change from pre-intervention (baseline) to post-intervention (30min later) on study day 1
  BOLD signal is used to measure the activity in the striatum as a predefined ROI, using Brainnetome atlas, following the delivery of aversive outcomes during 3-arm bandit task
Influence of abstinence duration on value coding | Change from pre-intervention (baseline) to post-intervention (60min later) on study day 1
  Across participants, correlation of number of days since last use of amphetamine with ∆BIC during contextual RL task
Influence of craving on value coding | Change from pre-intervention (baseline) to post-intervention (60min later) on study day 1
  Across participants, correlation of intensity of craving for amphetamine with ∆BIC during contextual RL task
Influence of withdrawal on value coding | Change from pre-intervention (baseline) to post-intervention (60min later) on study day 1
  Across participants, correlation of intensity of withdrawal for amphetamine with ∆BIC during contextual RL task

CONTACTS AND LOCATIONS:
Overall Officials: Maelle Gueguen, PhD, Principal Investigator — Laureate Institute for Brain Research, Inc.
Locations (1):
- Laureate Institute for Brain Research, Tulsa, Oklahoma, United States